CLINICAL TRIAL: NCT00537992
Title: Blue Light-Filter IOLs in Vitrectomy Combined With Cataract Surgery: Results of a Randomized Controlled Clinical Trial.
Brief Title: Blue-Blocking IOLs in Combined Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR-CI-03-2007
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Epiretinal Membranes; Macular Holes; Cataract
Keywords: combined surgery,; cataract surgery,; vitrectomy,; blue light-filter iols
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations; Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: combined surgery — UV-filter IOL (transparent IOL group) or a blue light-filter IOL (yellow IOL group) combined with a vitreoretinal procedure

SUMMARY:
Although commonly used in cataract surgery, the use of the blue light-filter IOLs in vitrectomy combined with cataract surgery has not been reported yet. A prospective controlled clinical trial was designed to evaluate the effect of the blue light-filter IOL on the surgeon's ability to perform specific vitreoretinal procedures and on the patients' outcome.

DETAILED DESCRIPTION:
Sixty patients were randomly assigned to receive a UV-filter IOL (transparent IOL group) or a blue light-filter IOL (yellow IOL group) combined with a vitreoretinal procedure.

Outcome measures were intraoperative conditions for the surgeon, complication rates, the functional outcome and vitreoretinal diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis vitreoretinal pathology (diabetic vitreous hemorrhage, macular hole, epiretinal membrane or persisting macula edema)
* Coexisting significant cataract
* The need for combined surgery ( pars plana vitrectomy, phacoemulsification and IOL implantation)
* Age over 50 years.

Exclusion Criteria:

* Pseudophakia on the non-study eye
* The need for silicone oil tamponade
* Optic atrophy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-10; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
intraoperative conditions for the surgeon (scaled questionnaire) and patients´ outcome

SECONDARY OUTCOMES:
complication rates and vitreoretinal diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, Prof., MD, Principal Investigator — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery; Christiane I Falkner-Radler, MD, Study Director — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery

REFERENCES:
- [Background] Hayashi K, Hayashi H. Visual function in patients with yellow tinted intraocular lenses compared with vision in patients with non-tinted intraocular lenses. Br J Ophthalmol. 2006 Aug;90(8):1019-23. doi: 10.1136/bjo.2006.090712. Epub 2006 Apr 5. PMID 16597662
- [Background] Olson RJ, Werner L, Mamalis N, Cionni R. New intraocular lens technology. Am J Ophthalmol. 2005 Oct;140(4):709-16. doi: 10.1016/j.ajo.2005.03.061. Epub 2005 Jul 18. PMID 16023990
- [Derived] Falkner-Radler CI, Benesch T, Binder S. Blue light-filter intraocular lenses in vitrectomy combined with cataract surgery: results of a randomized controlled clinical trial. Am J Ophthalmol. 2008 Mar;145(3):499-503. doi: 10.1016/j.ajo.2007.10.021. Epub 2008 Jan 11. PMID 18191090